CLINICAL TRIAL: NCT00222027
Title: GRAALL 2003 Trial (ALL 15-59 Years). Feasibility of Risk-Adapted Therapy in Young Adult Acute Lymphoblastic Leukemia: a Multicenter Trial
Brief Title: Feasibility of Risk-Adapted Therapy in Young Adult Acute Lymphoblastic Leukemia: a Multicenter Trial
Acronym: GRAALL2003
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: LLAU Marie-Elise, University Hospital Toulouse
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0200701; PHRC
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2009-01-07 (Estimated); Status verified 2009-01

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Acute lymphoblastic leukemia; adult patient; chemotherapy; stem cell transplantation; Young adult patients
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Collection of treatment-stratefying prognostic factors

SUMMARY:
Several prognostic predictors, including baseline ALL features and response to initial therapy, have been described in adult ALL raising the issue of whether these predictors might be redundant and which must be considered for treatment stratification. In the GRAALL-2003 prospective Phase 2 study, we aim to hierarchize the following high-risk factors in Ph-negative ALL patients.

DETAILED DESCRIPTION:
1) baseline (BL) : WBC30G/L in B-lineage, CNS involvement, MLL-AF4 and E2A-PBX fusions, haploidy/near-triploidy; 2) early response (ER) : corticoresistance after prophase (CsR), chemoresistance at Day 8 (ChR); all CsR and/or ChR patients are planned to receive higher doses of cyclophosphamide (HyperC) at Day 15 of induction; 3) induction response (IR) : no CR or Ig-TCR minimal residual disease (MRD) 10-2 after standard or HyperC induction. Allogeneic stem cell transplantation is proposed to patients with a donor and at least one BL, ER, or IR factor.

ELIGIBILITY:
Inclusion Criteria:

* 15-59 years
* acute lymphoblastic leukemia newly diagnosed
* signed written informed consent

Exclusion Criteria:

* Lymphoblastic lymphoma
* Acute lymphoblastic leukemia 3
* Chronic Myeloid Leukemia acutisation
* Sever organ condition

Ages: 15 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300
Dates: Start 2003-11; Primary Completion 2008-10 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Hierarchical evaluation of baseline poor-prognosis factors and response to initial therapy in younger adults with ALL

SECONDARY OUTCOMES:
Hematologic and non hematologic toxicity of induction, consolidation and late intensification.

CONTACTS AND LOCATIONS:
Overall Officials: Françoise HUGUET-RIGAL, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Service d'Hématologie Clinique, Hôpital Purpan, Toulouse, France

REFERENCES:
- [Derived] Delafoy M, Bonnet MF, Lengline E, Cieslak A, Touzart A, Balducci E, Simonin M, Lheritier V, Dourthe ME, Heid-Picard B, Latour S, Dombret H, Rousselot P, Baruchel A, Boissel N, Andrieu GP, Asnafi V. LEF1 intragenic deletion induces a dominant-negative isoform and unveils a Wnt/beta-catenin vulnerability in T-ALL. Blood. 2025 Dec 18;146(25):3036-3049. doi: 10.1182/blood.2025030161. PMID 40857670
- [Derived] Simonin M, Vasseur L, Lengline E, Lhermitte L, Cabannes-Hamy A, Balsat M, Schmidt A, Dourthe ME, Touzart A, Graux C, Grardel N, Cayuela JM, Arnoux I, Gandemer V, Huguet F, Ducassou S, Lheritier V, Chalandon Y, Ifrah N, Dombret H, Macintyre E, Petit A, Rousselot P, Lambert J, Baruchel A, Boissel N, Asnafi V. NGS-based stratification refines the risk stratification in T-ALL and identifies a very-high-risk subgroup of patients. Blood. 2024 Oct 10;144(15):1570-1580. doi: 10.1182/blood.2023023754. PMID 38848537
- [Derived] Balducci E, Simonin M, Duployez N, Steimle T, Dourthe ME, Villarese P, Ducassou S, Arnoux I, Cayuela JM, Balsat M, Courtois L, Andrieu G, Touzart A, Huguet F, Petit A, Ifrah N, Dombret H, Baruchel A, Macintyre E, Preudhomme C, Boissel N, Asnafi V. Genomic imbalance analysis provides new insight into prognostic factors in adult and pediatric T-ALL. Blood. 2024 Aug 29;144(9):988-1000. doi: 10.1182/blood.2023022154. PMID 38518104
- [Derived] Touzart A, Boissel N, Belhocine M, Smith C, Graux C, Latiri M, Lhermitte L, Mathieu EL, Huguet F, Lamant L, Ferrier P, Ifrah N, Macintyre E, Dombret H, Asnafi V, Spicuglia S. Low level CpG island promoter methylation predicts a poor outcome in adult T-cell acute lymphoblastic leukemia. Haematologica. 2020 Jun;105(6):1575-1581. doi: 10.3324/haematol.2019.223677. Epub 2019 Sep 19. PMID 31537687
- [Derived] Bond J, Touzart A, Lepretre S, Graux C, Bargetzi M, Lhermitte L, Hypolite G, Leguay T, Hicheri Y, Guillerm G, Bilger K, Lheritier V, Hunault M, Huguet F, Chalandon Y, Ifrah N, Macintyre E, Dombret H, Asnafi V, Boissel N. DNMT3A mutation is associated with increased age and adverse outcome in adult T-cell acute lymphoblastic leukemia. Haematologica. 2019 Aug;104(8):1617-1625. doi: 10.3324/haematol.2018.197848. Epub 2019 Jan 17. PMID 30655366
- [Derived] Bond J, Marchand T, Touzart A, Cieslak A, Trinquand A, Sutton L, Radford-Weiss I, Lhermitte L, Spicuglia S, Dombret H, Macintyre E, Ifrah N, Hamel JF, Asnafi V. An early thymic precursor phenotype predicts outcome exclusively in HOXA-overexpressing adult T-cell acute lymphoblastic leukemia: a Group for Research in Adult Acute Lymphoblastic Leukemia study. Haematologica. 2016 Jun;101(6):732-40. doi: 10.3324/haematol.2015.141218. Epub 2016 Mar 4. PMID 26944475
- [Derived] Chien WW, Catallo R, Chebel A, Baranger L, Thomas X, Bene MC, Gerland LM, Schmidt A, Beldjord K, Klein N, Escoffre-Barbe M, Leguay T, Huguet F, Larosa F, Hayette S, Plesa A, Ifrah N, Dombret H, Salles G, Chassevent A, Ffrench M. The p16(INK4A)/pRb pathway and telomerase activity define a subgroup of Ph+ adult Acute Lymphoblastic Leukemia associated with inferior outcome. Leuk Res. 2015 Apr;39(4):453-61. doi: 10.1016/j.leukres.2015.01.008. Epub 2015 Jan 25. PMID 25675863
- [Derived] Dhedin N, Huynh A, Maury S, Tabrizi R, Beldjord K, Asnafi V, Thomas X, Chevallier P, Nguyen S, Coiteux V, Bourhis JH, Hichri Y, Escoffre-Barbe M, Reman O, Graux C, Chalandon Y, Blaise D, Schanz U, Lheritier V, Cahn JY, Dombret H, Ifrah N; GRAALL group. Role of allogeneic stem cell transplantation in adult patients with Ph-negative acute lymphoblastic leukemia. Blood. 2015 Apr 16;125(16):2486-96; quiz 2586. doi: 10.1182/blood-2014-09-599894. Epub 2015 Jan 13. PMID 25587040
- [Derived] Beldjord K, Chevret S, Asnafi V, Huguet F, Boulland ML, Leguay T, Thomas X, Cayuela JM, Grardel N, Chalandon Y, Boissel N, Schaefer B, Delabesse E, Cave H, Chevallier P, Buzyn A, Fest T, Reman O, Vernant JP, Lheritier V, Bene MC, Lafage M, Macintyre E, Ifrah N, Dombret H; Group for Research on Adult Acute Lymphoblastic Leukemia (GRAALL). Oncogenetics and minimal residual disease are independent outcome predictors in adult patients with acute lymphoblastic leukemia. Blood. 2014 Jun 12;123(24):3739-49. doi: 10.1182/blood-2014-01-547695. Epub 2014 Apr 16. PMID 24740809
- [Derived] Trinquand A, Tanguy-Schmidt A, Ben Abdelali R, Lambert J, Beldjord K, Lengline E, De Gunzburg N, Payet-Bornet D, Lhermitte L, Mossafa H, Lheritier V, Bond J, Huguet F, Buzyn A, Leguay T, Cahn JY, Thomas X, Chalandon Y, Delannoy A, Bonmati C, Maury S, Nadel B, Macintyre E, Ifrah N, Dombret H, Asnafi V. Toward a NOTCH1/FBXW7/RAS/PTEN-based oncogenetic risk classification of adult T-cell acute lymphoblastic leukemia: a Group for Research in Adult Acute Lymphoblastic Leukemia study. J Clin Oncol. 2013 Dec 1;31(34):4333-42. doi: 10.1200/JCO.2012.48.5292. Epub 2013 Oct 28. PMID 24166518
- [Derived] Maury S, Huguet F, Leguay T, Lacombe F, Maynadie M, Girard S, de Labarthe A, Kuhlein E, Raffoux E, Thomas X, Chevallier P, Buzyn A, Delannoy A, Chalandon Y, Vernant JP, Rousselot P, Macintyre E, Ifrah N, Dombret H, Bene MC; Group for Research on Adult Acute Lymphoblastic Leukemia. Adverse prognostic significance of CD20 expression in adults with Philadelphia chromosome-negative B-cell precursor acute lymphoblastic leukemia. Haematologica. 2010 Feb;95(2):324-8. doi: 10.3324/haematol.2009.010306. Epub 2009 Sep 22. PMID 19773266